CLINICAL TRIAL: NCT02489435
Title: Randomized, Double-blind, Placebo-controlled, Phase Ib Clinical Trial of Safety and Pharmacokinetics of VM-1500 After Multiple Oral Administration in Healthy Volunteers
Brief Title: Clinical Trial of Safety and Pharmacokinetics of VM-1500 After Multiple Oral Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viriom (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02/HIV/2010
Record Dates: First submitted 2015-06-18; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-06

CONDITIONS: HIV-infection
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10 mg VM-1500 or Placebo (Experimental): VM-1500 for 9 volunteers, Placebo for 3 volunteers.
  Interventions: Drug: VM-1500; Drug: Placebo
- 20 mg VM-1500 or Placebo (Experimental): VM-1500 for 9 volunteers, Placebo for 3 volunteers.
  Interventions: Drug: VM-1500; Drug: Placebo
- 30 mg VM-1500 or Placebo (Experimental): VM-1500 for 9 volunteers, Placebo for 3 volunteers.
  Interventions: Drug: VM-1500; Drug: Placebo

INTERVENTIONS:
Drug: VM-1500 — VM-1500
Drug: Placebo — Placebo

SUMMARY:
The purpose of the study to assess safety and tolerability of VM-1500 and to determine main pharmacokinetic parameters of VM-1500 after multiple oral administration in adult healthy subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, phase Ib study in healthy volunteers with dose escalation to identify the optimal dosing schedule of VM-1500.

A total of 36 subjects will be treated with the VM-1500 or placebo for 14 days with further follow-up for four weeks. Subjects will be randomized into 3 cohorts with 3:1 drug/placebo ratio:

Cohort 1 (n=12): 10 mg VM-1500 for 9 volunteers, Placebo for 3 volunteers; Cohort 2 (n=12): 20 mg VM-1500 for 9 volunteers, Placebo for 3 volunteers; Cohort 3 (n=12): 30 mg VM-1500 for 9 volunteers, Placebo for 3 volunteers; Decision to escalate to the next (higher) dose will be made by the Independent Safety Review Board (ISRB), established specifically for this study. ISRB will base its decision on both the safety data obtained during drug administration in each cohort and analysis of clinical and lab data obtained within the course of the study.

Study time lines:

* Screening period - up to 30 days
* Treatment period - 14 days dosing (Day 1-14)
* 2 hospitalizations: Day 1-3, Day 13-15
* 28 PK samples in plasma: Day1 - predose, 0,25; 0,5; 1; 1,5; 2; 3; 4; 8; 12 hours Day 3, Day 5, Day 7, Day 9, Day 11, Day 13 - before dosing Day 14 (feed condition) - before dosing, 0,5; 1; 2; 4; 8; 12h Day 16, Day 23, Day 30, Day 37, Day 44 PK in blood cells - Day 1 (predose, 4h, 8h), Day 3, 5,7, 9, 11, 13, 14
* Post treatment follow-up period 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Provided signed written informed consent;
2. Healthy male subjects, 18-50 years of age;
3. Use of adequate and reliable forms of contraception during the study and 3 months after discontinuation of study medication.
4. ICF signed prior to any study-related procedure.

Exclusion Criteria:

1. HIV, hepatitis B, C antibodies in plasma;
2. Clinical relevant laboratory abnormalities;
3. Active tobacco, alcohol or drug abuse;
4. Anticipated non-compliance with the protocol;
5. Patients who have taken any investigational drug 3 months prior to the start of the study;
6. Plasma donorship, surgery 12 weeks prior to the start of the study;
7. Current significant gastrointestinal, renal, liver, bronchopulmonary, biliary, neurological, cardiovascular, oncologic, allergic, or ophthalmologic diseases, including history of cataracts/lens opacities.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of VM-1500 after multiple oral administration in adult healthy subjects based on analysis of AEs and laboratory values. | 14 days during drug administration plus follow-up for four weeks
Peak Plasma concentration (Cmax) of VM-1500 after multiple oral administration in adult healthy subjects. | 14 days during drug administration plus follow-up for four weeks
Area under the plasma concentration(AUC) of VM-1500 after multiple oral administration in adult healthy subjects. | 14 days during drug administration plus follow-up for four weeks
Plasma elimination half-life (T1/2) of VM-1500 after multiple oral administration in adult healthy subjects. | 14 days during drug administration plus follow-up for four weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Central Clinical City Hospital, Reutov, Moscow Oblast, Russia